CLINICAL TRIAL: NCT00186914
Title: Stromal Therapy of Osteodysplasia After Allogeneic Bone Marrow Transplantation: A Phase I Study
Brief Title: Stromal Therapy of Osteodysplasia After Allogeneic Bone Marrow Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Drexel University (Other); Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOD
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Osteodysplasia
Keywords: Bone marrow transplant; bone marrow stromal cells; allogeneic transplant; Osteodysplasia; Osteogenesis imperfecta; Gene marking; Stromal cell
MeSH Terms: conditions — Mucopolysaccharidosis IV; Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Biological: Marrow stromal cell infusion

INTERVENTIONS:
Biological: Marrow stromal cell infusion — This is a pilot study of infusions of ex vivo expanded, gene marked donor bone marrow stromal cells following allogeneic bone marrow transplantation. The study is a within patient dose escalation safety evaluation. It is believed that this patient population may benefit from these donor stromal cell infusions.
  As the stromal cells will be obtained from the original stem cell donor, no conditioning is required.
  Patients will receive two infusions of mesenchymal cells (MSC) approximately 14 to 21 days apart unless there is unacceptable toxicity after the first infusion. The first dose of cells to be given will be 1x10^6 MSC/kg and the second dose of cells will be 5x10^6 MSC/kg. The patients will be followed for approximately 28 days following the second infusion for any toxicity. Only after all six patients have safely completed both infusions will we consider 5 x 10^6 MSC/kg a safe dose of allogeneic mesenchymal stem cells for infusion.
  Other Names: Gene marking; mesenchymal cells

SUMMARY:
Osteodysplasia or poorly formed bones, "brittle bones" is a genetic disease with no known proven treatments. Some forms of osteodysplasia may cause severe disability and even death.

Eligible patients were limited to those children with Osteodysplasia who had undergone a previous allogeneic bone marrow transplant at St. Jude. The study intervention involved an infusion of a specified number of ex vivo expanded stromal cells obtained from the bone marrow of the same donor from whom they received their primary transplant procedure. These bone marrow stromal cells can become bone-forming cells, called osteoblasts. Participants then received 2 infusions of ex vivo expanded, gene marked cells not less than 6 months after bone marrow transplantation. The second cell infusion occurred between 14 to 21 days after the first infusion in the absence of toxicity. The goal of the study was to evaluate the safety and toxicity of these infusions.

DETAILED DESCRIPTION:
* To determine whether these ex vivo expanded, gene marked marrow stromal cells will engraft in the recipient's bone, bone marrow, and/or skin.
* To begin to investigate whether high proliferative mesenchymal progenitor cells can be expanded ex vivo and retain their progenitor potential in vivo.
* To begin to investigate whether ex vivo expanded bone marrow stromal cells can ameliorate the skeletal dysplasias associated with various genetic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an appropriate genetic disorder who have had an allogeneic bone marrow transplant and currently maintain complete or mixed hematopoietic chimerism
* Patient must be < or equal to 18Kg

Exclusion Criteria:

* Presence of infection
* Presence of GVHD (graft versus host disease)or the need for prophylaxis
* Concurrent participation in any investigational study that could potentially confound the interpretation of the safety parameters being investigated in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1999-07; Primary Completion 2001-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the stromal cell infusion | June 2001

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kasow, DO, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org